CLINICAL TRIAL: NCT00682708
Title: Sentinel Surveillance of Acute Malnutrition in the Region of Maradi, Niger, Children Under 5: Impact of a Preventive Intervention
Brief Title: Sentinel Surveillance of Malnutrition, Niger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Epicentre (Other)
Collaborators: Ministry of Health, Niger (Unknown); Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Rebecca Freeman Grais, epidemiologist, Epicentre
Purpose: Prevention
Other Study IDs: 07056
Record Dates: First submitted 2008-03-26; First posted 2008-05-22 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Malnutrition
Keywords: malnutrition; ready to use food; Niger
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: PlumpyNut
Dietary Supplement: PlumpyDoz

SUMMARY:
Malnutrition is a critical public health problem in developing countries. Malnutrition may be linked to more than one half of the deaths in children under 5 years old. In July 2001, after an intervention related to a measles epidemic, Medecins sans Frontieres-France opened a nutritional program in Maradi, in the South of Niger. The introduction of ready to use therapeutic foods (RUTF), in particular Plumpy'Nut (Nutriset, France) allowed for the treatment of the majority of children at their homes using ambulatory treatment. Children with complicated cases were cared for in an inpatient center. With ambulatory treatment the number of children cared for in the MSF program reached close to 70000 in 2006.

This study aimed to assess the effect of a 3-month distribution of RUTF in the context of a preventative supplementary feeding program. The primary hypotheses were that short-term RUTF supplementation at the village-level would prevent declines in weight-for-height and reduce the incidence of wasting in children 6 to 60 mo of age over a period of 8 mo. Because RUTF may have additional health effects, the intervention effect on height-for-age, stunting, mortality and morbidity from malaria, diarrhea, and respiratory infection were also examined.

ELIGIBILITY:
Inclusion Criteria:

* All children resident in randomized villages 6-59 months

Exclusion Criteria:

* N/A

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Start 2006-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
weight-for-height in children 6 to 60 mo of age | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca F Grais, Principal Investigator — Epicentre

REFERENCES:
- [Derived] Isanaka S, Nombela N, Djibo A, Poupard M, Van Beckhoven D, Gaboulaud V, Guerin PJ, Grais RF. Effect of preventive supplementation with ready-to-use therapeutic food on the nutritional status, mortality, and morbidity of children aged 6 to 60 months in Niger: a cluster randomized trial. JAMA. 2009 Jan 21;301(3):277-85. doi: 10.1001/jama.2008.1018. PMID 19155454